CLINICAL TRIAL: NCT02647021
Title: Evaluating Outcomes From a Combined Supervised Therapeutic and Physical Exercise Program for Post-surgical Head and Neck Cancer Survivors: A Randomized Controlled Trial
Brief Title: Therapeutic Resistance Group Exercise Training for Head & Neck Cancer Survivors
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Principal Investigator, Margie McNeely, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC.15-0167
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Neoplasms; Accessory Nerve Injury; Fatigue
Keywords: physical therapy; cancer rehabilitation; exercise
MeSH Terms: conditions — Head and Neck Neoplasms; Accessory Nerve Injuries; Fatigue; Motor Activity | interventions — Exercise Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Exercise (Active Comparator): Therapeutic Exercise Program (standard care) will include:
  1. Neck range of motion and strengthening, and posture retraining.
  2. Shoulder specific progressive resistance exercise program that focuses on spinal accessory nerve dysfunction and rehabilitation of trapezius muscle function.
  Interventions: Behavioral: Therapeutic Exercise
- Therapeutic + Lower Body Exercise (Experimental): The Therapeutic Exercise Program (standard care) will include:
  1. Neck range of motion and strengthening, and posture retraining.
  2. Shoulder specific progressive resistance exercise program that focuses on spinal accessory nerve dysfunction and rehabilitation of trapezius muscle function.
  The Resistance Exercise component will target 6-8 muscle groups of the lower extremities and core including gluteal, quadriceps, hamstrings, abdominals, and gastrocnemius muscles. A progressive introduction of exercises will occur over the first 3 weeks.
  1. a personalized program of lower extremity resistance exercises
  2. core strengthening exercises
  Interventions: Behavioral: Therapeutic Exercise; Behavioral: Therapeutic + Lower Body Exercise

INTERVENTIONS:
Behavioral: Therapeutic Exercise — A specialized therapeutic exercise program to address neck and shoulder dysfunction due to spinal accessory nerve damage.
Behavioral: Therapeutic + Lower Body Exercise — A combined therapeutic exercise program (as per the comparison arm) plus the addition of lower body resistance exercise
  Arms: Therapeutic + Lower Body Exercise

SUMMARY:
The investigators will conduct a randomized controlled trial examining 12-week, 24-week and one year outcomes from a combined therapeutic and physical exercise program that aims to bridge head-and-neck cancer survivors from acute care rehabilitation services to community-based exercise programming.

DETAILED DESCRIPTION:
Participants will be stratified by early (within 18 months of surgery) and late (> 18 months of surgery) and randomized on a one-on-one basis to (1) a supervised therapeutic exercise program for the neck and shoulder (serving as standard care) or (2) a combined therapeutic and lower body resistance exercise program. The randomization sequence will be generated by staff in the Rehabilitation Research Centre at Corbett Hall and placed in sealed opaque envelopes.

The exercise program will be offered in a group setting. Participants will exercise 2 times per week for a 10-week session and will have the option to continue for an additional 10-week maintenance session. The primary outcome for the study will be quality of life as measured by the Functional Assessment of Cancer Therapy (FACT)-Fatigue Scale at 12-weeks.

At each measurement point following the baseline assessment, including the 12-week and 24-week and one year follow-ups, an Independent Assessor will perform the objective fitness measurements. The Independent Assessor will also administer the Neck Dissection Impairment Questionnaire and the FACT-Fatigue quality of life questionnaires. The Physical Activity Adherence Diary will be collected by a Research Coordinator at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma/ thyroid cancer/ melanoma or lymphoma involving: oral cavity, oropharynx, larynx or hypopharynx, or lymph nodes in the neck region
* Surgical treatment includes radical neck dissection, modified radical neck dissection and other variants of functional/selective neck dissection OR radiation therapy to lymph node regions
* Presenting with shoulder and/ or neck dysfunction related to cancer treatment
* Karnofsky Performance Status greater than or equal to 60%
* No evidence of residual cancer in the neck and no distant (M0) metastasis. Potential participants with symptoms suggestive of distant metastasis (M1) must have appropriate investigations (e.g. bone scan) to rule these out.
* Participants must have completed their head and neck/ thyroid/ melanoma/ lymphoma cancer treatment (minimum 4 weeks post treatment)
* Pre-participation Screening: Prior to participation in the exercise program, potential participants will complete general and cancer-specific Physical Activity Readiness Questionnaires (PAR-Q+) to determine appropriateness for the exercise program. Physician consent and approval for supervised exercise will be required prior to enrollment.

Exclusion Criteria:

* A participant will be ineligible if they present with medical illness or psychiatric illness, which, in the opinion of the investigators, would impact his/her ability to participate in exercise or interfere with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy: Fatigue Scale Questionnaire | change from baseline to 12 weeks.
  Cancer related fatigue

SECONDARY OUTCOMES:
Shoulder range of motion in degrees. | Change from baseline to one year
  Active and passive glenohumeral joint range of motion using standard 12 inch goniometer.
Body mass index | Change from baseline to 24 weeks.
  Derived from height and weight of the participant.
1 repetition maximum (1RM) strength for seated row in pounds. | Change from baseline to 12 weeks.
  The maximal amount weight that can be pulled (seated row) and pushed (vertical bench) with proper form.
Neck Range of Motion in degrees. | Change from baseline to 12 weeks.
  Measures of neck flexion, side flexion, rotations and extension using myrin goniometer.
Upper extremity muscular endurance: number of repetitions performed. | baseline, 12-weeks, 24-weeks, one year
  Maximal repetitions to fatigue based on 50% of 1 repetition maximum strength for seated row.
Lower extremity flexibility in centimetres. | Change from baseline to 12-weeks.
  Sit and reach test
Functional capacity | Change from baseline to 24 weeks.
  6 minute walk test
Neck Dissection Impairment Index | Change from baseline to one year.
  Neck dissection related quality of life
Grip strength in pounds. | Change from baseline to 12-weeks.
  Maximal grip strength: composite score of both hands. Best of three attempts for each side.
1 repetition maximum leg press in pounds | Change from baseline to 12 weeks.
  The maximal amount of weight that can be moved with proper
1 repetition maximum chest press in pounds. | Change from baseline to 12 weeks.
  The maximal amount of weight that can be pushed with proper form.
30 second sit to stand (optional: in lieu of leg press) | Change from baseline to 12 weeks.
  number of repetitions performed in 30 seconds
Functional Assessment of Cancer Therapy Questionnaire Trial Outcome Index | Baseline to 12-weeks.
  The composite score of physical, functional and fatigue subscales of the questionnaire.

OTHER OUTCOMES:
Physical activity level in minutes per week (average over the previous one month period). | Change in monthly average physical activity from baseline to one year.
  Godin Leisure Time Questionnaire: minutes of mild, moderate and strenuous exercise.
Cost of programming | one year
  costs to programming, institution and participants
Exercise Adherence | Change from baseline to 1 year.
  Adherence to exercise programming: attendance at supervised exercise sessions and self-directed sessions over the 1 year period.
Functional Assessment of Cancer Therapy Fatigue Scale at one year. | Change from baseline to 1 year.
  Cancer-related fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. McNeely, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No